CLINICAL TRIAL: NCT06075082
Title: The Effect of the LEFT Smartwatch App as Sleep Positional Therapy for Nocturnal Gastroesophageal Reflux Symptoms.
Acronym: LEFT-APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. A.J. (Arjan) Bredenoord, Prof. dr. A.J. Bredenoord, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL83321.018.22
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Gastroesophageal Reflux; Heartburn
Keywords: Sleep positional therapy
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep positional therapy by using the LEFT smartwatch app (Experimental)
  Interventions: Device: LEFT smartwatch app

INTERVENTIONS:
Device: LEFT smartwatch app — The LEFT smartwatch app is an app on the Apple Watch which measures body sleep position and gently vibrates when the body is in the right lateral decubitus position. In this way, patients with nocturnal gastroesophageal reflux symptoms learn to avoid the right lateral sleep position as they will avoid the annoying vibrations. Measurements while using the smartwatch app will be compared to measurements at baseline.

SUMMARY:
The main objectives of the study are (1) to investigate if sleep positional therapy, using the LEFT smartwatch app reduces nocturnal gastroesophageal reflux symptoms in patients with gastroesophageal reflux disease symptomatology at night and (2) stimulates patients to avoid sleeping in the right lateral sleep position.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is one of the most common gastro-intestinal disorders and approximately 50-80% of the GERD patients experience nocturnal gastroesophageal reflux symptoms. Symptoms at night have a negative impact on sleep quality, daytime functioning and quality of life. When sleeping in left lateral decubitus position, the stomach is positioned below the esophagus, resulting in less reflux compared to sleeping in right lateral decubitus position. Sleep positional therapy, using an electronic wearable device which gently vibrates in an annoying way when turning in the sleep to the disadvantageous right lateral decubitus position, stimulates subjects to avoid sleeping in the right lateral decubitus position and effectively alleviates nocturnal gastroesophageal reflux symptoms. This prospective single center interventional pilot study will aim to (1) investigate if sleep positional therapy, using the LEFT smartwatch app reduces nocturnal gastroesophageal reflux symptoms in patients with GERD symptomatology at night and (2) stimulates patients to avoid sleeping in the right lateral sleep position.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Both male and female patients will be included.
* Age 18 years or older.
* Symptoms of heartburn and/or acid regurgitation during at least three nights a week.
* A total reflux symptom score ≥8 (measured through the GERDQ questionnaire score).
* Able to wear the Apple Watch on the left wrist.

Exclusion Criteria:

* Complete PPIs non-responders.
* Nightshift workers
* Surgery of the esophagus or stomach.
* Regular use of sleep medication (benzodiazepines) or medication which affect gastrointestinal motility (e.g. prokinetics or opioids) that cannot be stopped during the duration of the trial.
* Severe and clinically unstable concomitant disease (e.g. liver, cardiovascular or lung disease, neurological or psychiatric disorders, cancer or AIDS and other endocrine disorders)
* Patients with obstructive sleep apnea or esophageal motility disorders.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Nocturnal Gastroesophageal Reflux Disease Symptom Severity and Impact Questionnaire (N-GSSIQ) | 2 weeks
  The primary efficacy measure is relative change in total nocturnal gastroesophageal reflux symptoms measured by the Nocturnal Gastroesophageal Reflux Disease Symptom Severity and Impact Questionnaire (N-GSSIQ).
  The N-GSSIQ is a 20-item questionnaire measuring the severity, morning impact and concern about nocturnal gastro-esophageal reflux disease. The N-GSSIQ is a validated questionnaire to assess nocturnal GERD symptom severity over the past 2 weeks. The N-GSSIQ is comprised of three subscales: Nocturnal Gastroesophageal Reflux Disease Symptom Severity (13 questions, score range 0-65), Morning Impact of Nocturnal Gastroesophageal Reflux Disease (2 questions, score range 0-10), and Concern about Nocturnal Gastroesophageal Reflux Disease (5 questions, score range 0-20). Total score ranging from 0 to 95. A higher score indicates more severe symptoms.

SECONDARY OUTCOMES:
Treatment success | 2 weeks
  Percent responders as treatment success, defined as subjects with a minimal 50% reduction in nocturnal gastroesophageal reflux symptoms measured by N-GSSIQ
Change in total Nocturnal Gastroesophageal Reflux Disease Symptom Severity and Impact Questionnaire (N-GSSIQ) score. | 2 weeks
  Change in total Nocturnal Gastroesophageal Reflux Disease Symptom Severity and Impact Questionnaire (N-GSSIQ) score.
  The N-GSSIQ is a 20-item questionnaire measuring the severity, morning impact and concern about nocturnal gastro-esophageal reflux disease. The N-GSSIQ is a validated questionnaire to assess nocturnal GERD symptom severity over the past 2 weeks. The N-GSSIQ is comprised of three subscales: Nocturnal Gastroesophageal Reflux Disease Symptom Severity (13 questions, score range 0-65), Morning Impact of Nocturnal Gastroesophageal Reflux Disease (2 questions, score range 0-10), and Concern about Nocturnal Gastroesophageal Reflux Disease (5 questions, score range 0-20). Total score ranging from 0 to 95. A higher score indicates more severe symptoms.
Sleep position | 2 weeks
  Change in sleep position. Four sleep positions will be studied: left lateral decubitus, right lateral decubitus, supine and prone. The outcome sleep position will be noted as percentage of the time sleeping in a certain sleep position during the entire sleep.
Number of nocturnal reflux free nights | 2 weeks
  Change in the number of nocturnal reflux free nights measured by daily symptom diary
Reflux disease questionnaire (RDQ) | 2 weeks
  Change in reflux symptoms measured by Reflux disease questionnaire (RDQ) questionnaire.
  The RDQ is a validated 12-item questionnaire to obtain information on the current severity and frequency of reflux symptoms (heartburn, regurgitation and dyspepsia). The three subscales are the different reflux symptoms and consist of four questions. Scores were scaled with a Likert scale which ranges from 0 to 5. Subjects have more frequent and severe reflux symptoms if the RDQ score is higher
Pittsburgh Sleep Quality Index (PSQI) | 2 weeks
  Change in sleep quality measured by Pittsburgh Sleep Quality Index (PSQI).
  The PSQI is a validated 19-item questionnaire assessing various factors relating to sleep quality, sleep disturbance and usual sleep habits. The 19 items are grouped into seven component scores (sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction). The seven component scores are summed to calculate a global PSQI score, which has a range of 0-21. A higher score indicates a worse sleep quality; and a score above 5 is suspect for insomnia.
Functional Outcomes of Sleep Questionnaire (FOSQ) | 2 weeks
  Change in sleep quality measured by Functional Outcomes of Sleep Questionnaire (FOSQ).
  The FOSQ is a validated questionnaire about sleep-quality of life which consists of 30 questions. The short form which consists of 10 questions will be used in this study. Questions have a 4-point Likert scale. The recall period is not specified, but two weeks will be used in this study. A lowerscore indicates a worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands